CLINICAL TRIAL: NCT00492271
Title: A Double-Blind, Placebo-Controlled, Randomized, Dose-Escalating Study of Single (Part A) and Multiple (Part B) Intravenous Doses of Friulimicin B in Healthy Subjects
Brief Title: First Time in Man Trial for Friulimicin B
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unfavourable Pharmakokinetics
Sponsor: MerLion Pharmaceuticals GmbH (Industry)
Responsible Party: Michael Sieberling, MD; Principal Investigator, SWISS PHARMA CONTRACT LTD, Basel, Switzerland
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNB-001
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2008-07

CONDITIONS: Community Acquired Pneumonia; Staphylococcal Skin Infections
Keywords: Friulimicin B; Lipopeptide Antibiotic; First in Man
MeSH Terms: conditions — Community-Acquired Pneumonia; Staphylococcal Skin Infections | interventions — friulimicin B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Experimental arm with increasing dosage
  Interventions: Drug: Friulimicin B

INTERVENTIONS:
Drug: Friulimicin B — Intravenous, once daily, single dose

SUMMARY:
The purpose of this study is to study the safety of single doses and multiple doses of Friulimicin B in healthy volunteers. The level of Friulimicin B will be measured in the subjects blood and urine. One part of the study will assess if Friulimicin B in the plasma of subjects has activity against bacteria.

DETAILED DESCRIPTION:
Continued widespread use of antibiotics has promoted the spread of antibiotic resistance and has created an urgent need for antibacterial agents with no known cross resistance to other antibiotics available for humans. Friulimicin B has been shown to be highly active against a range of bacteria including such important pathogens such as methicillin resistant Staphylococcus aureus (MRSA), drug resistant Streptococcus pneumoniae and Glycopeptide resistant Enterococcus spp. These organisms are the causative agents in serious infections such as skin and soft tissue infections, pneumonia, bacteremia and endocarditis, complicated urinary tract infections, and osteomyelitis.

This study is the first use of Friulimicin B in man and will examine its safety and a preliminary study will assess if Friulimicin B in the plasma of subjects has activity against bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy subjects
* 18-55 years of age
* In good health

Exclusion Criteria:

* Abnormal physical findings of clinical significance at the Screening examination or baseline which would interfere with the objectives of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single and multiple intravenous doses of Friulimicin B by assessing adverse events, physical examinations,clinical chemistry examination, hematology, ECG and urinalysis. | 5 days

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of single and multiple intravenous doses of Friulimicin B in healthy subjects | 5 days
To determine the bactericidal activity of serum obtained from healthy subjects after administration of Friulimicin B | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sieberling, MD, Principal Investigator — Swiss Pharma Contract
Locations (1):
- Swiss Pharma Contract Ltd, Basel, Switzerland